CLINICAL TRIAL: NCT01762124
Title: Native Outflow Tract Transcatheter Pulmonary Valve Research Clinical Study
Brief Title: Study of the Native Outflow Tract Transcatheter Pulmonary Valve (TPV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Heart Valves (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 10022972DOC
Record Dates: First submitted 2012-11-30; First posted 2013-01-07 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Congenital Heart Disease; Tetralogy of Fallot
Keywords: Pulmonary valve; Congenital heart disease; Transcatheter pulmonary valve; Percutaneous pulmonary valve
MeSH Terms: conditions — Heart Defects, Congenital; Tetralogy of Fallot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Native Outflow Tract TPV (Experimental): Implantation of the Native Outflow Tract TPV
  Interventions: Device: Native Outflow Tract TPV

INTERVENTIONS:
Device: Native Outflow Tract TPV — Transcatheter placement of a pulmonary valve
  Other Names: Native TPV

SUMMARY:
The purpose of this early feasibility study is to determine how a new transcatheter pulmonary valve will move and perform once implanted in the right ventricular outflow tract.

DETAILED DESCRIPTION:
Medtronic, Inc. is in the process of developing a novel transcatheter device option for patients with congenital heart disease, without right ventricle-to-pulmonary artery conduits, called the Native Outflow Tract Transcatheter Pulmonary Valve. Given limitations in the animal model to confirm device boundary conditions, this feasibility study is proposed to characterize that information as well as evaluate safety, procedural feasibility and performance data to be used for future development of the device.

ELIGIBILITY:
Inclusion Criteria:

* Subject has pulmonary regurgitation as per one or more of the following criteria: Severe pulmonary regurgitation as measured by Doppler echocardiography, or Pulmonary regurgitant fraction ≥ 30% as measured by cardiac magnetic resonance imaging
* Clinical indication for surgical placement of a RVOT conduit or bioprosthetic pulmonary valve per one or more of the following criteria: Subject is symptomatic secondary to pulmonary insufficiency (e.g. exercise intolerance, fluid overload) as classified by the Investigator, or Right ventricular end diastolic volume (RVEDV) ≥ 150 ml/m2
* Subject is willing to consent to participate in the study and will commit to completion of all follow-up requirements

Exclusion Criteria:

* Anatomy unable to accommodate a 25 Fr delivery system
* Obstruction of the central veins
* Clinical or biological signs of infection including active endocarditis
* Indicated for intervention of stenosis of the branch pulmonary arteries at time of implant
* Positive pregnancy test at baseline (prior to CT angiography and again prior to implant procedure) in female subjects of child bearing potential
* Patients with right ventricular outflow tract obstruction (RVOTO) lesions surgically treated with a right ventricle-to-pulmonary artery conduit implant
* A major or progressive non-cardiac disease (e.g. liver failure, renal failure, cancer) that results in a life expectancy of less than one year
* Planned implantation of the Native Outflow Tract TPV in the left heart
* RVOT anatomy or morphology that is unfavorable for anchoring
* Known allergy to aspirin, heparin, or nickel
* Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
* Pre-existing prosthetic heart valve or prosthetic ring in any position
* Patient is currently enrolled in another investigational device or drug trial that may influence the outcome of this trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Measurement of radial, linear and axial compression, bending and torsion of device | 4 Days Post-Implant
  The following variables will be measured: radial compression, linear compression, axial compression, device bending and device torsion using the discharge CT. The degree of deformation of the device will be reported.

SECONDARY OUTCOMES:
Number of Patients with Procedural Success | 24 hours post-implant
  The number of patients who are successfully implanted with the device will be reported. This is measured by meeting all of the following criteria: Confirmation that the device is fixated within the desired location, RV-PA peak-to-peak gradient is less than 25 mmHg, Pulmonary regurgitation is moderate or less, and the subject is free of explantation at 24 hours post-implant.
Number of Patients with Serious Procedural Adverse Events | Through 5 year follow-up
  The number of patients that experience a serious procedural adverse event, as defined per the study protocol, will be reported.
Number of Patients with Device-related Adverse Events | Through 5 years
  The number of patients that experience a device-related adverse event, as defined per the study protocol, will be reported.
Number of Patients with Stent Fracture | Through 5 years
  The number of patients that experience a stent fracture of their device will be reported.
Number of Patients with Catheter Re-intervention on the TPV | Through 5 years
  The number of patients that experience a catheter re-intervention will be reported.
Assessment of Surgical Intervention on the TPV | Through 5 years
  The number of patients that undergo a surgical intervention will be reported.
Number of Patient Deaths (all-cause, procedural, and device-related) | Through 5 years
  Any patient deaths that occur during the study will be reported.
Pulmonary Regurgitant Fraction (%) as measured by cardiac MRI | Through 5 years
  The pulmonary regurgitant fraction for all patients, as measured by cardiac MRI, will be reported.
Pulmonary Regurgitation Severity as Measured by Echocardiography | Through 5 years
  The pulmonary regurgitation severity for all patients, as measured by echocardiography, will be reported.
Right Ventricular Volume (ml) as Measured by Cardiac MRI | Through 5 years
  The right ventricular volumes for all patients, as measured by cardiac MRI, will be reported.
Mean RVOT Gradient (mmHg) as Measured by Color Wave Doppler | Through 5 years
  The mean RVOT gradient for all patients, as measured by Color Wave Doppler, will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Benson, MD, Principal Investigator — The Hospital for Sick Children, Toronto, Canada; John P. Cheatham, MD, Principal Investigator — Nationwide Children's Hospital, Columbus, Ohio, USA; Lisa Bergersen, MD, MPH, Principal Investigator — Boston Children's Hospital, Boston, Massachusetts, USA
Locations (3):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Nationwide Children's Hospital, Columbus, Ohio
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morray BH, Gillespie MJ, Cheatham JP, Salavitabar A, Peng L, Jones TK, Levi DS, Gray RG, Asnes J, Cabalka AK, Fujimoto K, Qureshi AM, Bergersen L, Benson LN, Haugan D, McElhinney DB. Midterm Outcomes in a Pooled Cohort of Harmony Transcatheter Pulmonary Valve Recipients. Circ Cardiovasc Interv. 2025 Sep;18(9):e015196. doi: 10.1161/CIRCINTERVENTIONS.125.015196. Epub 2025 Jul 16. PMID 40665900
- [Derived] Gillespie MJ, Bergersen L, Benson LN, Weng S, Cheatham JP. 5-Year Outcomes From the Harmony Native Outflow Tract Early Feasibility Study. JACC Cardiovasc Interv. 2021 Apr 12;14(7):816-817. doi: 10.1016/j.jcin.2021.01.046. No abstract available. PMID 33826508
- [Derived] Benson LN, Gillespie MJ, Bergersen L, Cheatham SL, Hor KN, Horlick EM, Weng S, McHenry BT, Osten MD, Powell AJ, Cheatham JP. Three-Year Outcomes From the Harmony Native Outflow Tract Early Feasibility Study. Circ Cardiovasc Interv. 2020 Jan;13(1):e008320. doi: 10.1161/CIRCINTERVENTIONS.119.008320. Epub 2020 Jan 9. PMID 32525412